CLINICAL TRIAL: NCT00509574
Title: Association of Genetic Polymorphisms With Lipid Lowering Effects of Statin Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tzung-Dau Wang, MD, PhD, National Taiwan University Hospital
Other Study IDs: 200702006M
Record Dates: First submitted 2007-07-29; First posted 2007-07-31 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-11

CONDITIONS: Statins, HMG-CoA; Single Nucleotide Polymorphism
Keywords: Single Nucleotide Polymorphism; statins; hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples are obtained for genomic DNA extraction.
Oversight: Data Monitoring Committee: No

SUMMARY:
The 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors, also known as statins, played an important role in lipid-lowering therapy and reduction of cardiovascular risks. However, it has been observed that the response to statin therapy varies from patient to patient, and gene polymorphism could have contributed to the variation.

DETAILED DESCRIPTION:
Hyperlipidemic patients are retrospectively screened from 2006/1/1 to 2006/12/31. The patient is included if he or she had been receiving atorvastatin or rosuvastatin for at least 3 months and did not receive other lipid-lowering medications 4 weeks before starting atorvastatin or rosuvastatin. Genomic DNA was collected from the blood sample of each patient using genomic DNA purification kit. The single nucleotide polymorphisms (SNPs) were determined afterward.

The correlation between response of statin therapy, defined as changes in lipid profiles including triglyceride, total cholesterol, high density lipoprotein cholesterol and low density lipoprotein cholesterol, and SNPs examined.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-80.
* conforms with the criteria of National Cholesterol Education Program Adult Treatment Panel III for medication therapy.
* have received atorvastatin or rosuvastatin regularly for 12 weeks or longer.
* available lipid profiles such triglyceride, total cholesterol, high density lipoprotein cholesterol and low density lipoprotein cholesterol 12-24 weeks after staring statin therapy.

Exclusion Criteria:

* had been using lipid-lowering medications including statins 4 weeks before starting atorvastatin or rosuvastatin.
* received other lipid-lowering medications, erythromycin, immunosuppressant or azole antifungals concomitantly.
* pregnant, breast-feeding, or able to become pregnant.
* have a history of alcohol or substance abuse.
* liver cirrhosis or ALT exceeds the upper limit of normal range.
* untreated hypothyroidism.
* patients with malignant tumor who have received chemotherapy or radiotherapy.
* known allergy to atorvastatin, rosuvastatin or other statins.
* unwilling to provide written informed consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperlipidemic patients meeting the criteria of NCEP ATPIII for drug treatment at internal medicine clinic of National Taiwan University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-03; Study Completion 2010-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan